CLINICAL TRIAL: NCT03361332
Title: Behavioural and Neurofunctional Correlates of the Sense of Agency
Brief Title: The Sense of Agency
Acronym: SOA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: SOA
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Motor Activity; Motor Tic Disorders
MeSH Terms: conditions — Motor Activity; Tic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects
  Interventions: Other: Behavioral and fMRI
- Patients with Gilles de la Tourette Syndrome
  Interventions: Other: Behavioral and fMRI

INTERVENTIONS:
Other: Behavioral and fMRI — Subjects and patients will perform temporal-judgment-tasks (considered an indirect measure of the sense of agency) in an event-related fMRI setting. In the first task, they will hear a sound either caused by a voluntary key press or by the passive displacement of the same finger by the experimenter. Following each trial, subjects will estimate the delay between the finger movement and the subsequent sound, which will be presented at variable latencies after the key press. There will be also control-trials characterized by the active or passive movement with a subsequent sound presented with a delay that excludes causality inferences.

SUMMARY:
The ability to recognize of being the actors of the behaviour and its consequences, the so-called "Sense of Agency" (SoA), is a crucial component of self-awareness. One key aspect is the distinction from a mere inference about the causality between an act and its consequences and the sense of being the agent of it. Despite a large number of behavioural studies, there is unsatisfactory evidence on the functional anatomical underpinnings of the SoA and the distinction between causality and the SoA proper. Here, the investigators use an implicit measurement of the SoA and its modulations during fMRI: the intentional binding phenomenon (IB). The ivestigators also study how the SoA and the ensuing neurophysiological correlates are modulated by the presence of a movement disorders, such as Gilles de la Tourette Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age included between 18 and 65 years
* Right handed
* No contraindication to the fMRI exam

Exclusion Criteria:

* Contraindication to the fMRI exam

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy controls and patients with Gilles de la Tourette Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-04-08 (Actual); Primary Completion 2017-07-29 (Actual); Study Completion 2020-01-23 (Estimated)

PRIMARY OUTCOMES:
BOLD signal changes | April 2017 - October 2019
  The investigators will measure the changes of the BOLD signal associated with the modification of the sense of agency both in healthy subjects and neurological patients.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Galeazzi Orthopedic Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No